CLINICAL TRIAL: NCT01024699
Title: A Prospective Multi-Center Randomized Evaluation of the Clinical and Radiographic Outcomes of XLIF® Compared With MAS® TLIF for the Treatment of Symptomatic Lumbar Degenerative Spondylolisthesis With or Without Central Stenosis
Brief Title: XLIF® vs. MAS®TLIF for the Treatment of Symptomatic Lumbar Degenerative Spondylolisthesis With or Without Central Stenosis.
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.X0901
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- XLIF: This group will have the XLIF procedure done.
- MAS TLIF: This group will have the MAS TLIF procedure done.

SUMMARY:
The purpose of this study is to determine differences in the XLIF and TLIF procedures with respect to perioperative variables in adult patients with low-grade symptomatic spondylolisthesis.

DETAILED DESCRIPTION:
The study is a prospective multi-center randomized evaluation of clinical and radiographic outcomes of two commonly used lumbar interbody fusion procedures (XLIF and TLIF) in adult patients with low-grade symptomatic spondylolisthesis. The study seeks to identify differences between the procedures with respect to perioperative variables.

ELIGIBILITY:
Inclusion Criteria:

- Male and female patients who are at least 18 years of age;

- Patients who present with symptomatic Grade I or II degenerative spondylolisthesis at 1 or 2 contiguous lumbar levels between L1 and L5 and are surgical candidates for interbody lumbar fusion surgery; symptoms should include radiculopathy and/or neurogenic claudication with or without back pain;

- Patients who have been unresponsive to at least 6 months of conservative treatments or exhibit progressive neurological symptoms in the face of conservative treatment;

- Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the study.

Exclusion Criteria:

- Patients with lumbar pathologies requiring treatment at more than 2 levels;

- Patients who have had previous lumbar fusion surgery;

- Patients with lytic spondylolisthesis or a defect of the pars interarticularis;

- Patients with radiographic confirmation of Grade IV facet joint disease or degeneration;

- Patients with non-contained or extruded herniated nucleus pulposus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of patients from participating site locations.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The average improvement in clinical function (ODI) at 24 months compared with baseline, for each procedure. | 24 months

SECONDARY OUTCOMES:
The average improvement in pain (VAS) at 24 months compared with baseline, for each procedure. | 24 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - St. Vincent-Jacksonville, Jacksonville, Florida
  - Celebration Florida Hospital, Kissimmee, Florida
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - Northwest Orthopaedic Specialists, P.S., Paducah, Kentucky
  - Orthopaedic Clinic-Riverside Campus, University of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - The Methodist Hospital, Houston, Texas
  - Spine and Sports Institute, Richland, Washington
  - Northwest Orthopaedic Specialists, P.S., Spokane, Washington